CLINICAL TRIAL: NCT01935011
Title: Effects of the Stimulation Frequency of STN DBS on Swallowing Function in Patients With Parkinson's Disease
Brief Title: DBS Frequency on Swallowing Function in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0566
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PD DBS 60 Hz, 130 Hz or DBS off: PD DBS on 60 Hz stimulation, 130 Hz stimulation or DBS off
  Interventions: Other: PD, DBS

INTERVENTIONS:
Other: PD, DBS — PD DBS frequency on swallowing function

SUMMARY:
The stimulation frequency has been found to affect the axial symptoms of freezing of gait (FOG) and speech in advanced Parkinson's disease (PD) patients with subthalamic nucleus deep brain stimulation (STN DBS), with the traditionally high stimulation frequency of 130 Hz worsening while low frequency of 60 Hz improving these symptoms. The effect of stimulation frequency on another important axial symptom, swallowing dysfunction, has not been studied. The investigators hypothesize that stimulation frequency could have similar effect on swallowing function.

DETAILED DESCRIPTION:
This is the first study on the effect of the stimulation frequency on swallowing function in PD patients with STN DBS. Swallowing dysfunction is often difficult to treat pharmacologically and associated with increased morbidity and mortality. This study hence would have significant clinical implications in the management of swallowing dysfunction in these PD patients with STN DBS and could potentially decrease their morbidity and mortality.

The investigators expect that the traditionally high frequency stimulation of 130 Hz would worsen while the low frequency stimulation of 60 Hz would improve the swallowing function in OPMS summary

ELIGIBILITY:
Inclusion Criteria:

* Eight PD patients with STN DBS and freezing of gait responsive to stimulation frequency changes will be enrolled.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight PD patients with STN DBS and freezing of gait responsive to stimulation frequency changes will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome would be the OPMS swallowing function scores | One year
  Eight PD patients with STN DBS and FOG responsive to stimulation frequency changes will be enrolled. Information on the oropharyngeal motility study (OPMS) of the oral, pharyngeal and esophageal phase function will be collected, under "Med on/DBS off", "Med on/DBS 130 Hz", or "Med on/DBS 60 Hz". Each patient will be randomly assigned to these three conditions in a double blinded manner of 30 minutes apart. The patients will be reassessed under the single best condition (likely Med on/DBS 60 Hz) after being on for 6-8 weeks. ANOVA will be used for group comparison of the scores. A regression model will be further used to assess the predicting value (s) of the other scores and demographics for the swallowing function.

SECONDARY OUTCOMES:
The secondary outcome would be the swallowing questionnaire score | One year
  Eight PD patients with STN DBS and FOG responsive to stimulation frequency changes will be enrolled. Information on the swallowing questionnaire will be collected, under "Med on/DBS off", "Med on/DBS 130 Hz", or "Med on/DBS 60 Hz". Each patient will be randomly assigned to these three conditions in a double blinded manner of 30 minutes apart. The patients will be reassessed under the single best condition (likely Med on/DBS 60 Hz) after being on for 6-8 weeks.
The secondary outcome would also be the unified PD rating scale | One year
  Eight PD patients with STN DBS and FOG responsive to stimulation frequency changes will be enrolled. Information on the unified PD rating scale will be collected, under "Med on/DBS off", "Med on/DBS 130 Hz", or "Med on/DBS 60 Hz". Each patient will be randomly assigned to these three conditions in a double blinded manner of 30 minutes apart. The patients will be reassessed under the single best condition (likely Med on/DBS 60 Hz) after being on for 6-8 weeks.
The secondary outcome would be the FOG questionnaire score | One year
  Eight PD patients with STN DBS and FOG responsive to stimulation frequency changes will be enrolled. Information on the FOG questionnaire will be collected, under "Med on/DBS off", "Med on/DBS 130 Hz", or "Med on/DBS 60 Hz". Each patient will be randomly assigned to these three conditions in a double blinded manner of 30 minutes apart. The patients will be reassessed under the single best condition (likely Med on/DBS 60 Hz) after being on for 6-8 weeks.
The secondary outcome would be the standing-walking-sitting test score | One year
  Eight PD patients with STN DBS and FOG responsive to stimulation frequency changes will be enrolled. Information on the standing-walking-sitting test will be collected, under "Med on/DBS off", "Med on/DBS 130 Hz", or "Med on/DBS 60 Hz". Each patient will be randomly assigned to these three conditions in a double blinded manner of 30 minutes apart. The patients will be reassessed under the single best condition (likely Med on/DBS 60 Hz) after being on for 6-8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, MD PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States